CLINICAL TRIAL: NCT06441136
Title: Characterizing the Impact of Presbyphonia on Social Interaction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew R. Hoffman (Other)
Responsible Party: Sponsor-Investigator, Matthew R. Hoffman, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202307188
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-03

CONDITIONS: Presbyphonia
Keywords: voice therapy; aging voice; voice disorder; speech
MeSH Terms: conditions — Voice Disorders; Speech | interventions — Patient Health Questionnaire; Mental Status and Dementia Tests; Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phonation Resistance Training Exercises (PhoRTE) Voice Therapy Program (Experimental): PhoRTE is a voice therapy program administered by a speech language pathologist for participants with presbyphonia. During sessions, participants perform five vocal exercises at individualized target vocal intensity. Goals of therapy are to increase muscular workload on vocal mechanism and target the respiratory and laryngeal muscular deficits that result from aging. Participants practice 6 days per week at home and meet with speech pathologist weekly for 4 weeks.
  Interventions: Other: PhoRTE Program; Other: University of California Los Angeles (UCLA) Loneliness Scale; Other: Social Disconnectedness Scale; Other: Patient Health Questionnaire 9; Other: Aging Voice Index; Other: The Edmonton Frail Scale; Other: Vocal Effort Scale; Other: Montreal Cognitive Assessment; Other: Voice Handicap Index-10; Other: Voice Problem Impact Scales; Other: Cough Severity Index; Procedure: Laryngoscopy; Other: Acoustic, perceptual, and aerodynamic assessments

INTERVENTIONS:
Other: PhoRTE Program — Speech therapy program guided by a speech language pathologist. This program includes in person or virtual visits and at home exercises.
  Other Names: Speech Therapy Program
Other: University of California Los Angeles (UCLA) Loneliness Scale — A questionnaire measuring levels of loneliness.
  Other Names: UCLA Loneliness Scale
Other: Social Disconnectedness Scale — A questionnaire that asks about social network size and the frequency of social activities attended.
Other: Patient Health Questionnaire 9 — A questionnaire measuring levels of depression.
  Other Names: PHQ-9
Other: Aging Voice Index — A questionnaire of patient-reported voice outcome measures designed to capture the quality of life impact of dysphonia in older adults.
Other: The Edmonton Frail Scale — A questionnaire that measures frailty levels.
Other: Vocal Effort Scale — A picture based questionnaire scale that asks the subject to rate their perceived effort when using their voice.
Other: Montreal Cognitive Assessment — A screening tool used to test for cognitive impairment.
  Other Names: MOCA
Other: Voice Handicap Index-10 — A questionnaire used to measure quality of life impact of dysphonia.
  Other Names: VHI-10
Other: Voice Problem Impact Scales — A 4 question survey that captures impact of voice on four domains - work/daily activities, social life, home, and overall quality of life.
  Other Names: VPIS
Other: Cough Severity Index — A 10 question survey asking to rate severity of cough.
Procedure: Laryngoscopy — Nose is anesthetized and a flexible endoscope is passed to visualize the larynx at rest and during sustained vowel production (/i/) for 3-5 seconds. This will be used to measure bowing index and normalized glottal gap of the vocal folds.
  Other Names: Flexible transnasal videostroboscopy
Other: Acoustic, perceptual, and aerodynamic assessments — Participants will complete voice recording tasks including sustained vowel production, six standard sentences, and 20 seconds of natural conversational speech. This will be used to measure CAPE-V rating, Cepstral peak prominence, fundamental frequency, signal-to-noise ratio, voice type components, mean flow rate, subglottal pressure, and vocal efficiency.

SUMMARY:
The purpose of this study is to determine if presbyphonia, or voice disorder caused by age-related change in the larynx, is associated with change in social interaction. This proposal investigates the impact of voice impairment in older adults on social interaction, loneliness, social disconnectedness, and depression. A series of questionnaires, voice assessments, and interviews will be performed to improve our understanding of how voice disorders affect older adults and how treatment of voice impairment with voice therapy may improve quality of life.

DETAILED DESCRIPTION:
During the study visit, all subjects (including the control group) will be given ten questionnaires asking them to rate their loneliness and quality of life in relation to the changes in their voice. All participants will undergo audiometry to assess hearing (with hearing aids if used at home). If they do not pass the hearing test, they will be screened out of the study.

Participants will then provide a required voice sample using sustained vowels for 3-5 seconds 5 times each, repeating six standard sentences, and 20 seconds of natural conversational speech. Using this voice recording, the following assessments and measurements will be obtained: CAPE-V rating (Consensus auditory perceptual evaluation of voice), Cepstral peak prominence (measurement of dysphonia), fundamental frequency, signal-to-noise ratio, and voice type components (captures breathiness).

Subjects will then be asked to produce a train of /pi pi pi/ at a comfortable pitch and loudness into a mask with an intra-oral mouthpiece to record both pressure and airflow. Five trials will be performed. The following measurements will be obtained: mean flow rate, subglottal pressure, and vocal efficiency.

Subjects will then undergo an awake videostroboscopy using a small flexible camera passed through the nose to view the vocal folds. During this procedure, the nose is anesthetized and the subject is asked to produce sustained vowels for 3-5 seconds. This part of the study takes about 2 minutes to complete. The parameters to be measured for this are: bowing index of the vocal folds and normalized glottal gap.

For the second part of this study, subjects from the presbyphonia population only will be recruited to participate in the phonation resistance training exercises or PhoRTE voice therapy. Prior to therapy, for two weeks, participants will take pictures when their voice disorder may be affecting them or ability to socialize. Brief journal entry will be completed. Photos will be collected, printed, and used as memory recall tool for a pre-treatment semi-structured interview. Interviews will be conducted, approximately 45-60 minutes induration. Both online and in-person options will be available to facilitate participation. An interview guide will include questions designed to assess participants' perception of voice and how voice affects social participation.

Subjects will then complete PhoRTE therapy. Participants perform 5 vocal exercises at individualized target vocal intensity. Goals of therapy are to increase muscular workload on vocal mechanism and target the respiratory and laryngeal muscular deficits that result from aging. Participants practice 6 days per week at home and meet with speech pathologist weekly for 4 weeks.

Following therapy, participants will participate in 60-75-minute semi-structured small group interviews approximately 3 months after voice therapy. Interviews will address experience with voice therapy, and any changes after voice therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of presbyphonia with findings of presbylaryngis on videostroboscopy, with findings of bilateral true vocal fold atrophy and normal vocal fold motion bilaterally
* Able to complete all questionnaires and voice assessment tasks
* Normal to mild hearing loss in aided condition (with hearing aids)

Exclusion Criteria:

* Liquid dysphagia or pneumonia in the last year
* Vocal fold lesion/scar/motion impairment
* Neurologic disorder affecting the voice
* Montreal cognitive assessment score <26 or <25 if 12 or fewer years of formal education

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The Effect on Loneliness with the PhoRTE Voice Therapy Program | Baseline and at 3 months
  Loneliness will be measured using the University of California - Los Angeles (UCLA) Loneliness Scale questionnaire at baseline and at the end of the 4-week PhoRTE program. The UCLA Loneliness Scale is a 20-item scale with each item rated on a 4-point Likert scale (ranging from 1, "never," to 4, "often") and the total score can range from 20 to 80, with higher scores indicating greater feelings of loneliness.

SECONDARY OUTCOMES:
The Effect on Social Disconnectedness with the PhoRTE Voice Therapy Program | Baseline and at 3 months
  Social disconnectedness will be measured using the Social Disconnectedness Scale questionnaire at baseline and at the end of the 4 week PhoRTE program. The Social Disconnectedness Scale is based on a 15-item scale with each item rated on their own scale depending on the question asked (ex: ranging from 0, "never" to 7, "several times a week" or indicating number of individuals in a social network). The total score can range from 2 to 72, with lower scores indicating greater levels of social disconnectedness.
The Effect on Depression with the PhoRTE Voice Therapy Program | Baseline and at 3 months
  Levels of depression will be measured using the Patient Health Questionnaire-9 (PHQ-9) at baseline and at the end of the 4 week PhoRTE program. The PHQ-9 is a 9-item scale with each item rated on a scale (ranging from 0, "not at all," to 3, "nearly every day") and the total score can range from 0-27 with higher scores indicating greater feelings of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Hoffman, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data or resources, shared upon request, will be de-identified and released only after appropriate data sharing agreements are completed by the relevant parties. Users must agree to the conditions of use governing access to the public release data. This includes restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, proper acknowledgement of the data resource, information provided to users will not be used for commercial purposes, and will not be redistributed to third parties.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after study completion
Access Criteria: email principal investigator
  a non-disclosure and/or data usage agreement will most likely be required

REFERENCES:
- [Background] Awan SN, Roy N, Dromey C. Estimating dysphonia severity in continuous speech: application of a multi-parameter spectral/cepstral model. Clin Linguist Phon. 2009 Nov;23(11):825-41. doi: 10.3109/02699200903242988. PMID 19891523
- [Background] Baertsch HC, Bhatt NK, Giliberto JP, Dixon C, Merati AL, Sauder C. Quantification of Vocal Fold Atrophy in Age-Related and Parkinson's Disease-Related Vocal Atrophy. Laryngoscope. 2023 Jun;133(6):1462-1469. doi: 10.1002/lary.30394. Epub 2022 Sep 16. PMID 36111826
- [Background] Baker TA, Wang CC. Photovoice: use of a participatory action research method to explore the chronic pain experience in older adults. Qual Health Res. 2006 Dec;16(10):1405-13. doi: 10.1177/1049732306294118. PMID 17079801
- [Background] Belsky MA, Rothenberger SD, Gillespie AI, Gartner-Schmidt JL. Do Phonatory Aerodynamic and Acoustic Measures in Connected Speech Differ Between Vocally Healthy Adults and Patients Diagnosed with Muscle Tension Dysphonia? J Voice. 2021 Jul;35(4):663.e1-663.e7. doi: 10.1016/j.jvoice.2019.12.019. Epub 2020 Jan 10. PMID 31932188
- [Background] Belsky MA, Shelly S, Rothenberger SD, Ziegler A, Hoffman B, Hapner ER, Gartner-Schmidt JL, Gillespie AI. Phonation Resistance Training Exercises (PhoRTE) With and Without Expiratory Muscle Strength Training (EMST) For Patients With Presbyphonia: A Noninferiority Randomized Clinical Trial. J Voice. 2023 May;37(3):398-409. doi: 10.1016/j.jvoice.2021.02.015. Epub 2021 Mar 16. PMID 33741235
- [Background] Cacioppo JT, Hughes ME, Waite LJ, Hawkley LC, Thisted RA. Loneliness as a specific risk factor for depressive symptoms: cross-sectional and longitudinal analyses. Psychol Aging. 2006 Mar;21(1):140-51. doi: 10.1037/0882-7974.21.1.140. PMID 16594799
- [Background] Catalani C, Minkler M. Photovoice: a review of the literature in health and public health. Health Educ Behav. 2010 Jun;37(3):424-51. doi: 10.1177/1090198109342084. Epub 2009 Oct 1. PMID 19797541
- [Background] Chan AW, Chan HY, Chan IK, Cheung BY, Lee DT. An Age-Friendly Living Environment as Seen by Chinese Older Adults: A "Photovoice" Study. Int J Environ Res Public Health. 2016 Sep 13;13(9):913. doi: 10.3390/ijerph13090913. PMID 27649217
- [Background] Cohen SM. Self-reported impact of dysphonia in a primary care population: an epidemiological study. Laryngoscope. 2010 Oct;120(10):2022-32. doi: 10.1002/lary.21058. PMID 20830762
- [Background] Cornwell EY, Waite LJ. Social disconnectedness, perceived isolation, and health among older adults. J Health Soc Behav. 2009 Mar;50(1):31-48. doi: 10.1177/002214650905000103. PMID 19413133
- [Background] Etter NM, Hapner ER, Barkmeier-Kraemer JM, Gartner-Schmidt JL, Dressler EV, Stemple JC. Aging Voice Index (AVI): Reliability and Validity of a Voice Quality of Life Scale for Older Adults. J Voice. 2019 Sep;33(5):807.e7-807.e12. doi: 10.1016/j.jvoice.2018.04.006. Epub 2018 May 7. PMID 29748025
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Gilman M, Merati AL, Klein AM, Hapner ER, Johns MM. Performer's attitudes toward seeking health care for voice issues: understanding the barriers. J Voice. 2009 Mar;23(2):225-8. doi: 10.1016/j.jvoice.2007.08.003. Epub 2007 Nov 26. PMID 18037270
- [Background] Giua R, Pedone C, Scarlata S, Carrozzo I, Rossi FF, Valiani V, Incalzi RA. Relationship between respiratory muscle strength and physical performance in elderly hospitalized patients. Rejuvenation Res. 2014 Aug;17(4):366-71. doi: 10.1089/rej.2014.1549. PMID 24749768
- [Background] Golub JS, Chen PH, Otto KJ, Hapner E, Johns MM 3rd. Prevalence of perceived dysphonia in a geriatric population. J Am Geriatr Soc. 2006 Nov;54(11):1736-9. doi: 10.1111/j.1532-5415.2006.00915.x. PMID 17087701
- [Background] Hartman DE. The perceptual identity and characteristics of aging in normal male adult speakers. J Commun Disord. 1979 Feb;12(1):53-61. doi: 10.1016/0021-9924(79)90021-2. PMID 422747
- [Background] Heman-Ackah YD, Sataloff RT, Laureyns G, Lurie D, Michael DD, Heuer R, Rubin A, Eller R, Chandran S, Abaza M, Lyons K, Divi V, Lott J, Johnson J, Hillenbrand J. Quantifying the cepstral peak prominence, a measure of dysphonia. J Voice. 2014 Nov;28(6):783-8. doi: 10.1016/j.jvoice.2014.05.005. Epub 2014 Aug 29. PMID 25179777
- [Background] Hennink M, Kaiser BN. Sample sizes for saturation in qualitative research: A systematic review of empirical tests. Soc Sci Med. 2022 Jan;292:114523. doi: 10.1016/j.socscimed.2021.114523. Epub 2021 Nov 2. PMID 34785096
- [Background] Holaday LW, Oladele CR, Miller SM, Duenas MI, Roy B, Ross JS. Loneliness, sadness, and feelings of social disconnection in older adults during the COVID-19 pandemic. J Am Geriatr Soc. 2022 Feb;70(2):329-340. doi: 10.1111/jgs.17599. Epub 2021 Dec 10. PMID 34850379
- [Background] Honjo I, Isshiki N. Laryngoscopic and voice characteristics of aged persons. Arch Otolaryngol. 1980 Mar;106(3):149-50. doi: 10.1001/archotol.1980.00790270013003. PMID 7356434
- [Background] House JS. Social isolation kills, but how and why? Psychosom Med. 2001 Mar-Apr;63(2):273-4. doi: 10.1097/00006842-200103000-00011. No abstract available. PMID 11292275
- [Background] Kaneko H, Suzuki A, Horie J. Relationship of Cough Strength to Respiratory Function, Physical Performance, and Physical Activity in Older Adults. Respir Care. 2019 Jul;64(7):828-834. doi: 10.4187/respcare.06490. Epub 2019 Feb 5. PMID 30723166
- [Background] Kim ME, Sund LT, Morton M, Kim J, Choi JS, Castro ME. Provider and Patient Satisfaction with Telemedicine Voice Therapy During the COVID-19 Pandemic. J Voice. 2025 Jan;39(1):282.e19-282.e27. doi: 10.1016/j.jvoice.2022.07.009. Epub 2022 Jul 18. PMID 36038478
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lin FC, Chien HY, Chen SH, Kao YC, Cheng PW, Wang CT. Voice Therapy for Benign Voice Disorders in the Elderly: A Randomized Controlled Trial Comparing Telepractice and Conventional Face-to-Face Therapy. J Speech Lang Hear Res. 2020 Jul 20;63(7):2132-2140. doi: 10.1044/2020_JSLHR-19-00364. Epub 2020 Jun 24. PMID 32579859
- [Background] Lindstrom E, Ohlund Wistbacka G, Lotvall A, Rydell R, Lyberg Ahlander V. How older adults relate to their own voices: a qualitative study of subjective experiences of the aging voice. Logoped Phoniatr Vocol. 2023 Dec;48(4):163-171. doi: 10.1080/14015439.2022.2056243. Epub 2022 Apr 21. PMID 35446741
- [Background] Liu B, Hao G, Cui Y, Fang J, Ji M, Wu J, Jiang J, Shao J, Liu H. Introduction of Voice Type Component (VTC) as an Effective Acoustic Voice Analysis Method in Tele-evaluation. J Voice. 2025 Nov;39(6):1463-1472. doi: 10.1016/j.jvoice.2023.07.005. Epub 2023 Aug 4. PMID 37544815
- [Background] Liu B, Polce E, Raj H, Jiang J. Quantification of Voice Type Components Present in Human Phonation Using a Modified Diffusive Chaos Technique. Ann Otol Rhinol Laryngol. 2019 Oct;128(10):921-931. doi: 10.1177/0003489419848451. Epub 2019 May 14. PMID 31084359
- [Background] Lockett D, Willis A, Edwards N. Through seniors' eyes: an exploratory qualitative study to identify environmental barriers to and facilitators of walking. Can J Nurs Res. 2005 Sep;37(3):48-65. PMID 16268089
- [Background] Ma EP, Yiu EM. Voice activity and participation profile: assessing the impact of voice disorders on daily activities. J Speech Lang Hear Res. 2001 Jun;44(3):511-24. doi: 10.1044/1092-4388(2001/040). PMID 11407557
- [Background] Marmor S, Horvath KJ, Lim KO, Misono S. Voice problems and depression among adults in the United States. Laryngoscope. 2016 Aug;126(8):1859-64. doi: 10.1002/lary.25819. Epub 2015 Dec 21. PMID 26691195
- [Background] Mau T, Jacobson BH, Garrett CG. Factors associated with voice therapy outcomes in the treatment of presbyphonia. Laryngoscope. 2010 Jun;120(6):1181-7. doi: 10.1002/lary.20890. PMID 20513037
- [Background] Mezzedimi C, Di Francesco M, Livi W, Spinosi MC, De Felice C. Objective Evaluation of Presbyphonia: Spectroacoustic Study on 142 Patients with Praat. J Voice. 2017 Mar;31(2):257.e25-257.e32. doi: 10.1016/j.jvoice.2016.05.022. Epub 2016 Jul 15. PMID 27427181
- [Background] Mund M, Maes M, Drewke PM, Gutzeit A, Jaki I, Qualter P. Would the Real Loneliness Please Stand Up? The Validity of Loneliness Scores and the Reliability of Single-Item Scores. Assessment. 2023 Jun;30(4):1226-1248. doi: 10.1177/10731911221077227. Epub 2022 Mar 4. PMID 35246009
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Mysyuk Y, Huisman M. Older people's emotional connections with their physical urban environment, Cities & Health, 2020; 4:1, 25-30.
- [Background] Novek Sheila, Morris-Oswald Toni, Menec Verena. Using photovoice with older adults: some methodological strengths and issues. Ageing & Society. 2012;32(3):451-470.
- [Background] Pessin AB, Tavares EL, Gramuglia AC, de Carvalho LR, Martins RH. Voice and ageing: clinical, endoscopic and acoustic investigation. Clin Otolaryngol. 2017 Apr;42(2):330-335. doi: 10.1111/coa.12725. Epub 2016 Sep 6. PMID 27537269
- [Background] Prince MJ, Harwood RH, Blizard RA, Thomas A, Mann AH. Social support deficits, loneliness and life events as risk factors for depression in old age. The Gospel Oak Project VI. Psychol Med. 1997 Mar;27(2):323-32. doi: 10.1017/s0033291796004485. PMID 9089825
- [Background] Radloff, L. S. The CES-D Scale: A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement. 1977; 1(3), 385-401.
- [Background] Rolfson DB, Majumdar SR, Tsuyuki RT, Tahir A, Rockwood K. Validity and reliability of the Edmonton Frail Scale. Age Ageing. 2006 Sep;35(5):526-9. doi: 10.1093/ageing/afl041. Epub 2006 Jun 6. No abstract available. PMID 16757522
- [Background] Rosen CA, Lee AS, Osborne J, Zullo T, Murry T. Development and validation of the voice handicap index-10. Laryngoscope. 2004 Sep;114(9):1549-56. doi: 10.1097/00005537-200409000-00009. PMID 15475780
- [Background] Roy N, Merrill RM, Gray SD, Smith EM. Voice disorders in the general population: prevalence, risk factors, and occupational impact. Laryngoscope. 2005 Nov;115(11):1988-95. doi: 10.1097/01.mlg.0000179174.32345.41. PMID 16319611
- [Background] Roy N, Stemple J, Merrill RM, Thomas L. Epidemiology of voice disorders in the elderly: preliminary findings. Laryngoscope. 2007 Apr;117(4):628-33. doi: 10.1097/MLG.0b013e3180306da1. PMID 17429872
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Samlan RA, Black MA, Abidov M, Mohler J, Fain M. Frailty Syndrome, Cognition, and Dysphonia in the Elderly. J Voice. 2020 Jan;34(1):160.e15-160.e23. doi: 10.1016/j.jvoice.2018.06.001. Epub 2018 Jul 25. PMID 30055984
- [Background] Shembel AC, Rosen CA, Zullo TG, Gartner-Schmidt JL. Development and validation of the cough severity index: a severity index for chronic cough related to the upper airway. Laryngoscope. 2013 Aug;123(8):1931-6. doi: 10.1002/lary.23916. Epub 2013 Jun 4. PMID 23737389
- [Background] Sillanpaa E, Stenroth L, Bijlsma AY, Rantanen T, McPhee JS, Maden-Wilkinson TM, Jones DA, Narici MV, Gapeyeva H, Paasuke M, Barnouin Y, Hogrel JY, Butler-Browne GS, Meskers CG, Maier AB, Tormakangas T, Sipila S. Associations between muscle strength, spirometric pulmonary function and mobility in healthy older adults. Age (Dordr). 2014;36(4):9667. doi: 10.1007/s11357-014-9667-7. Epub 2014 Jul 30. PMID 25073451
- [Background] Smith E, Verdolini K, Gray S, et al. Effect of voice disorders on quality of life. J Med Speech-Lang Path 1996; 4:223-44.
- [Background] Sprecher A, Olszewski A, Jiang JJ, Zhang Y. Updating signal typing in voice: addition of type 4 signals. J Acoust Soc Am. 2010 Jun;127(6):3710-16. doi: 10.1121/1.3397477. PMID 20550269
- [Background] Steffick, D. E. Documentation of affective functioning measures in the Health and Retirement Study (Tech. Rep. No. HRS/AHEAD). Ann Arbor, MI: Survey Research Center, University of Michigan. 2000; Available from http://hrsonline.isr.umich.edu/docs/userg/dr-005.pdf.
- [Background] Stek ML, Vinkers DJ, Gussekloo J, Beekman AT, van der Mast RC, Westendorp RG. Is depression in old age fatal only when people feel lonely? Am J Psychiatry. 2005 Jan;162(1):178-80. doi: 10.1176/appi.ajp.162.1.178. PMID 15625218
- [Background] Sundholm N, Shelly S, Wright ML, Reynolds J, Slovarp L, Gillespie AI. Effect of Behavioral Cough Suppression Therapy Delivered via Telehealth. J Voice. 2025 May;39(3):851.e1-851.e5. doi: 10.1016/j.jvoice.2022.11.015. Epub 2022 Dec 20. PMID 36550001
- [Background] Tenforde AS, Borgstrom H, Polich G, Steere H, Davis IS, Cotton K, O'Donnell M, Silver JK. Outpatient Physical, Occupational, and Speech Therapy Synchronous Telemedicine: A Survey Study of Patient Satisfaction with Virtual Visits During the COVID-19 Pandemic. Am J Phys Med Rehabil. 2020 Nov;99(11):977-981. doi: 10.1097/PHM.0000000000001571. PMID 32804713
- [Background] Timmons Sund L, Collum JA, Bhatt NK, Hapner ER. VHI-10 Scores in a Treatment-Seeking Population With Dysphonia. J Voice. 2023 Mar;37(2):290.e1-290.e6. doi: 10.1016/j.jvoice.2020.12.017. Epub 2021 Jan 13. PMID 33451893
- [Background] Titze I.R., ''Workshop on Acoustic Voice Analysis: Summary Statement,'' in Notional Center for Voice and Speech, CO: Denver, 1995, pp. 26-27.
- [Background] Vaca M, Mora E, Cobeta I. The Aging Voice: Influence of Respiratory and Laryngeal Changes. Otolaryngol Head Neck Surg. 2015 Sep;153(3):409-13. doi: 10.1177/0194599815592373. Epub 2015 Jul 8. PMID 26156424
- [Background] van Beljouw IMJ, van Exel E, de Jong Gierveld J, Comijs HC, Heerings M, Stek ML, van Marwijk HWJ. "Being all alone makes me sad": loneliness in older adults with depressive symptoms. Int Psychogeriatr. 2014 Sep;26(9):1541-1551. doi: 10.1017/S1041610214000581. PMID 24717770
- [Background] Verdonck-de Leeuw IM, Mahieu HF. Vocal aging and the impact on daily life: a longitudinal study. J Voice. 2004 Jun;18(2):193-202. doi: 10.1016/j.jvoice.2003.10.002. PMID 15193652
- [Background] Wang C, Burris MA. Photovoice: concept, methodology, and use for participatory needs assessment. Health Educ Behav. 1997 Jun;24(3):369-87. doi: 10.1177/109019819702400309. PMID 9158980
- [Background] Wang LH, Doan TN, Chang FC, To TL, Ho WC, Chou LW. Prevalence of Voice Disorders in Older Adults: A Systematic Review and Meta-Analysis. Am J Speech Lang Pathol. 2023 Jul 10;32(4):1758-1769. doi: 10.1044/2023_AJSLP-22-00393. Epub 2023 Jun 7. PMID 37285381
- [Background] Wilson JA, Deary IJ, Millar A, Mackenzie K. The quality of life impact of dysphonia. Clin Otolaryngol Allied Sci. 2002 Jun;27(3):179-82. doi: 10.1046/j.1365-2273.2002.00559.x. PMID 12071993
- [Background] Ziegler A, Verdolini Abbott K, Johns M, Klein A, Hapner ER. Preliminary data on two voice therapy interventions in the treatment of presbyphonia. Laryngoscope. 2014 Aug;124(8):1869-76. doi: 10.1002/lary.24548. Epub 2014 Jan 29. PMID 24375313